CLINICAL TRIAL: NCT04994600
Title: Design and Validation of a German Language Questionnaire for Measuring Alarm Fatigue in Nurses and Medical Doctors in Intensive Care Units
Brief Title: Design and Validation of a German Language Questionnaire for Measuring Alarm Fatigue in Intensive Care Units
Acronym: alarmZen1
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Vivantes Klinikum im Friedrichshain, Klinik für Anästhesie, Intensivmedizin, Notfallmedizin und Schmerztherapie, Landsberger Allee 49, 10249 Berlin (Unknown); Universitätsklinikum Gießen, UKGM GmbH, Justus-Liebig-Universität Gießen, Klinik für Anästhesiologie, Rudolf-Buchheim Str. 7, 35392 Gießen (Unknown); Universitätsklinikum Heidelberg, Klinik für Anästhesiologie, Im Neuenheimer Feld 420, 69120 Heidelberg (Unknown); Universitätsklinikum Ulm, Klinik für Anästhesiologie und Intensivmedizin, Albert-Einstein-Allee 23, 89081 Ulm (Unknown); Technische Universität München, Klinik für Anästhesiologie und Intensivmedizin, Klinikum rechts der Isar Ismaninger Str. 22, 81675 München (Unknown); Marien Hospital Herne, Universitätsklinikum der Ruhr-Universität Bochum Klinik für Anästhesiologie, Hölkeskampring 40, 44625 Herne (Unknown)
Responsible Party: Principal Investigator, Felix Balzer, Prof. Dr. med. Dr. rer. nat., Charite University, Berlin, Germany
Other Study IDs: alarmZen1
Record Dates: First submitted 2021-08-03; First posted 2021-08-06 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Alarm Fatigue
MeSH Terms: conditions — Alert Fatigue, Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EFA_1st_phase: Exploratory factor analysis group. All staff members (physicians, specialist nurses, respiratory therapists) of Charite intensive care units
- CFA_2nd_phase: Confirmatory factor analysis group. All staff members (physicians, specialist nurses, respiratory therapists) of collaborating intensive care units.
  Interventions: Other: Reduces number of question items

INTERVENTIONS:
Other: Reduces number of question items — The number of alarm fatigue questions are reduced to about 15 in the CFA_2nd_phase group.
  Groups: CFA_2nd_phase

SUMMARY:
False-positive and non-actionable alarms can lead to staff desensitization ("alarm fatigue") and thus patient endangerment. With this study the investigators create a basic tool to survey alarm fatigue of intensive care staff: the first German language alarm fatigue questionnaire.

DETAILED DESCRIPTION:
In intensive care units (ICUs), patients' vital signs are monitored automatically. As soon as one of the parameters indicates a critical or potentially critical condition, an alarm is triggered on the ward. However, if there are too many alarms, even most of which are false or require no treatment, ward staff may develop alarm fatigue and become desensitized to alarms. This puts patients at risk, especially by overhearing critical alarms. Overburdening staff with alarms is part of everyday life in most ICUs. Considering the demographic development as well as the COVID-19 pandemic, it is to be expected that the number of intensive care patients and thus also the alarm burden in intensive care units will increase. This will also be exacerbated by the increasing digitization of the ICU. Evidence-based and data-driven alarm management enables clinicians to trust alarms again. With this study the investigators create a basic tool to survey alarm fatigue of intensive care staff: the first German language alarm fatigue questionnaire. The questionnaire will be collected in two phases. With the data from the first phase (N ≈ 300), the investigators aim to uncover any structure that may be latent in the questionnaire data (by exploratory factor analysis) and reduce the number of questions from 27 to ~15. The reduced questionnaire will be collected in the second phase (N ≈ 300 - 400). With the data obtained, the investigators intend to test the structure postulated in the first survey in a confirmatory factor analysis.

ELIGIBILITY:
Inclusion Criteria:

* physicians of German intensive care units
* specialist nurses of German intensive care units
* respiratory therapists of German intensive care units

Exclusion Criteria:

- Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All staff members (physicians, specialist nurses, respiratory therapists) of German intensive care units.
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of alarm fatigue | 6 months
  Develop an online alarm fatigue survey questionnaire to be completed across campuses and hospitals by ICU staff.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Balzer, Prof. Dr. Dr., Principal Investigator — Charite Universitaetsmedizin Berlin
Locations (1):
- Charite Universtitaetsmedizin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided